CLINICAL TRIAL: NCT05179161
Title: Validation of Prone Crawl Radiotherapy for Whole-breast Irradiation After Breast Conserving Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC-UZ-2016/0351; B670201628048 (Registry Identifier: Belgian Registration Number)
Record Dates: First submitted 2021-10-19; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer Female
Keywords: Prone positioning; Prone crawl position; Radiotherapy; Whole breast irradiation; Setup errors; Patient comfort; Setup time; Deep inspiration breathhold; Dosimetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prone crawl position (Experimental): Patients are placed in the prone crawl position for whole breast irradiation and are treated with 15 x 2,67 Gy (± boost treatment if required as per international guidelines)
  Interventions: Device: Prone crawl positioning

INTERVENTIONS:
Device: Prone crawl positioning — Breast cancer patients are placed in a prone position with the ipsilateral arm besides the body rather than extended besides the head on a dedicated couch that provides the required support for maintaining this position.

SUMMARY:
The aim of this study is to validate the obtained results of setup precision, comfort and setup time. The possibility of using breath hold for heart sparing in combination with prone crawl position will be tested. Forty patients (20 with left-sided and 20 with right-sided breast carcinoma) presenting for WBI without LNI after breast-conserving surgery will be included after signing informed consent.

DETAILED DESCRIPTION:
This is a phase II non-randomized trial, where 40 patients will be treated for breast cancer requiring whole breast irradiation as per standard of care. Patients will be simulated and treated using the novel prone crawl position to a total dose of 40.05 Gy in 15 fractions of 2.67 Gy.

The trial aims to evaluate setup precision, patient comfort and setup time in the prone crawl positioning. Feasibility of deep inspiration breathhold will be tested and dosimetric parameters evaluated.

This is done through registration of setup errors at the time of treatment, questionnaires for comfort/discomfort scoring, time registration, toxicity scoring, and dosimetric analysis in treatment planning systems.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Non-metastasized breast carcinoma
* Multidisciplinary decision of adjuvant radiotherapy after lumpectomy for breast cancer
* Prone WBI without LNI indicated according to the department's guidelines, treatment schedule of at least 15 fractions
* Age ≥ 18 years
* Informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* < 18 years old
* Mastectomy
* Need for LNI
* Bilateral breast irradiation
* Partial breast irradiation
* Unable to be treated in prone position
* Less than 15 treatment fractions planned
* Situs inversus
* Pregnant or breastfeeding
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Setup error | During the intervention
  Setup errors are analyzed using Van Herk parameters obtained by rigid coregistration of treatment imaging with simulation imaging

SECONDARY OUTCOMES:
Patient comfort | immediately after the intervention
  Patient comfort as assessed by questionnaire
Setup Time | During the intervention
  Time taken for setting up the patient for each fraction
Reproducibility of DIBH | At baseline
  The reproducibility and stability of deep inspiration breathhold is investigated by performing multiple breathhold manoevres during CT imaging at baseline, and comparing the relative geometric position of organs between on the acquired images for each patient. This will be evaluated by calculating the overlap index and dice similarity coefficien between these images.
Acute toxicity | 6 months after treatment end
  Acute side effects due to radiotherapy using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 toxicity scoring system, scoring toxicities from grade 0 (no toxicity) to grade 5 (death)
Dose to target and dose to organs at risk | Before treatment initiation after CT simulation
  Analysis is dose using the Dose-volume histogram (DVH) of targets and organs at risk, as obtained on CT simulation images. These DVH's are used to assess amount of radiation received by each organ and treatment target and assess the risk of treatment failure or treatment harm.

CONTACTS AND LOCATIONS:
Overall Officials: Liv Veldeman, MD, PhD, Principal Investigator — University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No
Sharing patient data is not planned

REFERENCES:
- [Result] Deseyne P, Speleers B, De Neve W, Boute B, Paelinck L, Vakaet V, Van Hulle H, Schoepen M, Stouthandel M, Van Greveling A, Post G, Detand J, Monten C, Depypere H, Veldeman L. Crawl positioning improves set-up precision and patient comfort in prone whole breast irradiation. Sci Rep. 2020 Oct 2;10(1):16376. doi: 10.1038/s41598-020-72702-3. PMID 33009448
- [Derived] Deseyne P, Speleers B, Paelinck L, De Gersem W, De Neve W, Schoepen M, Van Greveling A, Van Hulle H, Vakaet V, Post G, Monten C, Depypere H, Veldeman L. Reproducibility of repeated breathhold and impact of breathhold failure in whole breast and regional nodal irradiation in prone crawl position. Sci Rep. 2022 Feb 3;12(1):1887. doi: 10.1038/s41598-022-05957-7. PMID 35115610